CLINICAL TRIAL: NCT06047834
Title: A Phase 2, Open-Label, Randomized, Controlled, Dose Cohort, Pharmacokinetic and Safety Study of Oral Lofexidine in Neonates Experiencing Opioid Withdrawal Due to Intrauterine Exposure to Opioids
Brief Title: Pharmacokinetic and Safety Study of Oral Lofexidine in Neonates Experiencing Opioid Withdrawal Due to Intrauterine Exposure to Opioids
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioCorRx Pharmaceuticals Inc (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USWM-LX2-2001
Record Dates: First submitted 2023-07-18; First posted 2023-09-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Opioid Withdrawal (Disorder)
MeSH Terms: interventions — Standard of Care; lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (Placebo Comparator): All participants will receive non pharmacologic interventions per the local standard of care (i.e. non-pharmacologic measures and morphine when indicated).
  Interventions: Other: Standard of Care without Lofexidine
- Dose 1 (Experimental): Drug: Lofexidine (LX2) All participants will receive standard of care and 32 µg/kg/day of Lofexidine, administered as 4 µg/kg/day every 3 hours. Lofexidine will be tapered to discontinuation.
  Interventions: Drug: Standard of Care with Lofexidine
- Dose 2 (Experimental): Drug: Lofexidine (LX2) All participants will receive standard of care and 20 µg/kg/day of Lofexidine, administered as 5 µg/kg/day every 3 hours. Lofexidine will be tapered to discontinuation.
  Interventions: Drug: Standard of Care with Lofexidine
- Dose 3 (Experimental): Drug: Lofexidine (LX2) All participants will receive standard of care and 16-24 µg/kg/day of Lofexidine, administered every 6 hours, with the final daily dose level to be decided based upon data collected in participants receiving Dose 2. Lofexidine will be tapered to discontinuation.
  Interventions: Drug: Standard of Care with Lofexidine

INTERVENTIONS:
Drug: Standard of Care with Lofexidine — Participants will be randomized 3:1 to treatment with standard of care with or without lofexidine. Subjects randomized to standard of care with lofexidine will be sequentially assigned to 1 of 3 dose levels: Dose 1 (32 μg/kg/day, administered as 4 μg/kg/day q3h), Dose 2 (20 μg/kg/day, administered as 5 μg/kg/day q6h), or Dose 3 (16 μg/kg/day to 24 μg/kg/day administered q6h, with the final daily dose level to be decided based on data collected in participants receiving Dose 2).
  Arms: Dose 1; Dose 2; Dose 3
Other: Standard of Care without Lofexidine — Participants will be randomized 3:1 to treatment with standard of care with or without lofexidine. Subjects randomized to standard of care without lofexidine wilt receive non-pharmacologic measures and morphine when indicated.
  Arms: Control

SUMMARY:
A randomized, open-label, controlled, ascending dose cohort, PK, and safety study assessing standard of care (i.e., non-pharmacologic measures and morphine when indicated) with or without lofexidine for the treatment of opioid withdrawal symptoms in neonates due to intrauterine exposure to opioids, described as neonatal opioid withdrawal syndrome (NOWS) or neonatal abstinence syndrome (NAS).

This study has been designed to assess the pharmacokinetics (PK) and safety of the lofexidine in neonates experiencing NOWS. The effectiveness of lofexidine on the severity of NOWS will also be evaluated. Results from this study will be used to support dosing recommendations in neonates and to inform further studies in the pediatric patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient's parent or legally authorized representative(s) (LAR)/guardian(s) in accordance with local laws and Institutional Review Board (IRB) requirements.
2. Infants <7 days of age at the time of randomization.
3. Gestational age ≥35 weeks at birth.
4. Minimum weight ≥1.8 kg at birth.
5. Infant's mother is ≥18 years of age.
6. Intrauterine opiate exposure expected to contribute to NOWS symptoms, as determined by the Principal Investigator and supported by at least one of the following:

   1. Maternal history of opiate use during pregnancy as confirmed by diagnosis of opioid use disorder (OUD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), treatment for OUD, treatment with an opioid prescribed by a licensed physician or health care worker, documentation of opiate use in maternal medical record, and/or maternal self-reported opiate use;
   2. Positive maternal urine opiate screen during pregnancy or delivery; or
   3. Participant urine, meconium, or cord blood or tissue testing positive for opiate metabolites.
7. Symptomatic with 2 consecutive scores ≥8 on the mFNAST at sites using the mFNAST OR at least one score ≥1 on the ESC assessment and with agreement from the clinical care team at sites using the ESC approach to care. Note: The study team should use the same NOWS scoring method (i.e., mFNAST or ESC assessment) to determine the patient's eligibility as is used to assess NOWS symptoms per the local standard of care.
8. Can receive medications orally.

Exclusion Criteria:

1. Patients who developed NOWS due to prolonged neonatal intensive care unit (NICU) analgesia and sedation therapy.
2. Received treatment for NOWS, including morphine, methadone, buprenorphine, clonidine, or phenobarbital before screening/randomization.
3. Prenatal exposure to an investigational drug, device, or biological agent other than investigational formulations of buprenorphine or methadone administered as part of treatment for maternal opioid dependence.
4. Any anticipated or scheduled surgery during the patient's inpatient treatment for NOWS through approximately 30 days after completion of their treatment for NOWS (not including circumcision).
5. Seizures, confirmed by EEG.
6. mFNAST score ≥14.
7. Two consecutive blood pressure measurements greater than 15 minutes apart with a systolic blood pressure <55 mm Hg.
8. Two consecutive heart rate measurements <110 bpm more than 15 minutes apart.
9. Clinically significant abnormal ECG at Screening in the judgment of the Principal Investigator, including a QTc interval >480 msec on a Screening ECG. Note: if the QTc interval meets the above criteria, the value may be confirmed by repeating the measurement twice, with each ECG obtained approximately 30-60 minutes apart, and the QTc interval confirmed by a pediatric cardiologist. If the pediatric cardiologist confirms the QTc interval is >480 msec based on two of the three ECGs, the patient will be excluded from participation. If the pediatric cardiologist confirms the QTc interval is ≤480 msec based on two of the three ECGs, the patient may be considered for study entry at the discretion of the Investigator in consultation with the pediatric cardiologist. Patients with a confirmed QTc >480 msec at Screening will be monitored per local standard of care, at least once daily, until the QTc resolves to within normal range. Patients not enrolled in the study will receive additional evaluation and care as clinically indicated.
10. Have clinically significant abnormal laboratory values on laboratory tests completed for clinical reasons, including laboratory values outside the normal range as determined by the local lab that would put the patient at undue risk, as determined by the Principal Investigator, including either of the following:

    1. Hematocrit values of <40%
    2. Platelet count <100,000/μL
11. Requiring sustained treatment with IV fluids or supplemental oxygen. Note: Patients with a transient need for IV fluids or supplemental oxygen may be considered for inclusion in the study at the Investigator's discretion.
12. Any congenital malformations or acute medical illness, condition, or clinical finding that, in the opinion of the Principal Investigator and/or the Sponsor, would put the patient at undue risk for study participation or interfere with the patient's ability to complete the study, including concerns related to medication administration or patient survival.

Ages: 0 Hours to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations following single dose and repeated lofexidine administration in participants | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution

SECONDARY OUTCOMES:
Single dose and steady-state maximum concentrations | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution
Extent of accumulation (i.e., Accumulation Ratio [AR]) with repeated dosing | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution
Examination of dose proportionality | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution
Estimation of apparent clearance | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution
Estimation of apparent volume of distribution | Day 1 through Day 7
  To evaluate the pharmacokinetic (PK) parameters of lofexidine granules for reconstitution
Treatment emergent adverse events (TEAEs) | Day 1 through 30 day follow-up
  To evaluate the safety of lofexidine during administration in infants experiencing NOWS

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall Health, Huntington, West Virginia, United States